CLINICAL TRIAL: NCT05002088
Title: Retrospective Assessment of the Portico Transcatheter Aortic Valve for Valve-in-Valve Use
Brief Title: Portico Valve-in-Valve Retrospective Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABBOTT-CIP-10414
Record Dates: First submitted 2021-07-27; First posted 2021-08-12 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Failure; Aortic Insufficiency; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Primary Analysis Population: The primary analysis population will include patients who have signed an Informed Consent Form, and at minimum, the Portico delivery system entered his/her vasculature for an attempted Portico ViV implant. Patients must have met the sizing requirements of the PorticoTM transthoracic aortic valve sizing specification (≥19 mm and ≤27 mm).
  Interventions: Device: Transcatheter Aortic Valve Replacement
- Exploratory Registry Arm: The exploratory registry arm will collect data for patients that were treated for a failed surgical bioprosthetic aortic valve true inner diameter size of <19 mm or >27 mm.
  Interventions: Device: Transcatheter Aortic Valve Replacement

INTERVENTIONS:
Device: Transcatheter Aortic Valve Replacement — Transcatheter Aortic Valve Replacement for the treatment of a failed surgical aortic valve bioprosthesis, Valve-in-Valve (ViV), in patients who were considered to be at increased risk for redo surgical aortic valve replacement

SUMMARY:
The objective of this data-collection study is to retrospectively evaluate the safety and clinical performance of the Portico transthoracic aortic valve for Valve-in-Valve treatment of a failed aortic surgical bioprosthetic valve in patients who are considered at increased surgical risk for a redo surgical aortic valve replacement.

DETAILED DESCRIPTION:
Two options currently exist to treat failed surgical aortic bioprostheses: transcatheter valve-in-valve implantation (ViV) or redo surgical aortic valve replacement (rAVR). The objective of this comprehensive data-collection study is to retrospectively evaluate the safety and clinical performance of the Portico transthoracic aortic valve for Valve-in-Valve treatment of a failed aortic surgical bioprosthetic valve in patients who are considered at increased surgical risk for a redo surgical aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Subject had a degenerated surgical aortic bioprosthetic valve with severe aortic stenosis, severe regurgitation, or a combination of at least moderate stenosis with at least moderate regurgitation per EAPCI-ESC-EACTS standardized criteria.
2. Surgical bioprosthesis true inner diameter (true ID) was ≥ 19 mm and ≤ 27 mm and was confirmed by either CT or confirmed by the Valve in Valve Aortic App. Refer to the PCR website https://www.pcronline.com/PCR-Publications/PCR-mobile-apps/Valve-in-Valve-Aortic-app Note: if CT was contraindicated and/or not possible to be obtained, a transesophageal echocardiogram (TEE) will be accepted for sizing.
3. Prior to Portico ViV procedure, the patient was deemed at increased risk for surgery to replace the surgical aortic bioprosthetic valve.
4. Subject provided written informed consent prior to performing data collection for study specific visits. For patients that are deceased at the time of enrollment, all institutional/local legal and regulatory requirements for consent must be met prior to enrollment and data collection.
5. Subject is ≥ 18 years of age or legal age in host country at the time of consent.
6. Prior to the Portico ViV index procedure, the subject had New York Heart Association (NYHA) class II, III, or IV.
7. Subject had a minimum vessel diameter of 6.0 mm for Portico™ delivery system access or a minimum of 5.0 mm for the FlexNav™ delivery system.
8. Subject had the Portico or FlexNav delivery system enter their vasculature

Exclusion Criteria:

1. Subject had evidence of an acute MI, percutaneous intervention, or a peripheral intervention ≤30 days prior to Portico ViV index procedure (MI defined as: ST Segment Elevation as evidenced on 12 Lead ECG).
2. Subject had uncontrolled blood dyscrasias defined as: leukopenia (WBC<3,000 mm3), acute anemia (Hb <9 g/dL), or thrombocytopenia (platelet count <50,000 cells/mm³).
3. Subject was considered hemodynamically unstable at the time of the ViV procedure (requiring inotropic support or mechanical heart assistance)
4. Subject had severe ventricular dysfunction with left ventricular ejection fraction (LVEF) <20% as measured by resting echocardiogram.
5. Subject had imaging evidence of intracardiac mass, thrombus or vegetation.
6. Subject had an active peptic ulcer or has/had upper gastrointestinal (GI) bleeding ≤3 months prior to ViV index procedure.
7. Subject had a documented history of a cerebrovascular accident (CVA) or a transient ischemic attack (TIA) ≤6 months prior to index procedure.
8. Subject had renal insufficiency (serum creatinine >3.0 mg/dL (265.5μmol/L)) and/or end stage renal disease requiring chronic dialysis.
9. Subject had active bacterial endocarditis or ongoing sepsis ≤ 6 months prior to the index procedure.
10. Surgical aortic bioprosthetic valve was unstable or rocking.
11. Subject had a vascular condition (i.e. stenosis, tortuosity, or severe calcification) that made insertion and endovascular access to the aortic valve impossible.
12. Subject was unable to tolerate antiplatelet or anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study may enroll up to 100 patients who had a documented failed surgical aortic bioprosthetic valve (due stenosis, insufficiency, or a combination of both) at increased risk for redo surgical aortic valve replacement surgery. Patients must have met the sizing requirements of the Portico transthoracic aortic valve sizing specification (≥19 mm and ≤27 mm). Patients must meet all inclusion and exclusion criteria to be eligible for enrollment.
  In addition, an exploratory registry arm will collect data for patients that were treated for a failed surgical bioprosthetic aortic valve true inner diameter size of <19 mm or >27 mm. There will be no enrollment limit in the exploratory registry arm
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, Study Director — Abbott
Locations (7):
- Australia (2):
  - GenesisCare - St Andrew's Hospital & GenesisCare Leabrook - Satellite Site of GenesisCare - Wesley Hospital, Adelaide
  - GenesisCare - Wesley Hospital, Auchenflower
- Rigshospitalet, Copenhagen, Denmark
- Germany (2):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Universitätsklinikum Rostock (AöR), Rostock
- United Kingdom (2):
  - St. Bartholomew's Hospital, London
  - Morriston Hospital - ABM University Health Board, Morriston

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 6 clinical sites from four countries enrolled a total of 71 subjects between October, 2021 and September, 2023. Subjects were enrolled to two cohorts: the Primary Cohort enrolled subjects with a surgical bioprosthesis true inner diameter (ID) between 19 mm and 27 mm, while the Exploratory Cohort enrolled subjects with a true ID outside that range.
  Once enrolled, subjects completed follow up visits at 30 days, 1-year, and annually through five years.
Period: Overall Study
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Started | 57 | 14
Completed | 7 | 4
Not Completed | 50 | 10
Not completed — Withdrawal by Subject | 9 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 16 | 2
Not completed — Protocol Violation | 25 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Analysis Population | Exploratory Registry Arm | Total
Number analyzed (Participants) | 57 | 14 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The age for one subject not available.
  years
    number analyzed (Participants) | 56 | 14 | 70
    (all) | 79.7 (6.2) | 80.6 (9.3) | 79.9 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 41 | 3 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 57 | 14 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 46 | 6 | 52
Ejection Fraction [Mean (Standard Deviation); unit: percent (%)] | 56.1 (10.2) | 59.5 (9.9) | 56.7 (0)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: The Rate of All-cause Mortality, Disabling Stroke, Life-threatening Bleeding Requiring Blood Transfusion, Acute Kidney Injury (AKI) Requiring Dialysis, and Major Vascular Complication.
Description: Composite of all-cause mortality, disabling stroke, life threatening bleeding requiring blood transfusion, acute kidney injury (AKI) requiring dialysis, and major vascular complications
Time Frame: 30 days post index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
Participants | 2 | 0

2. Primary Outcome: Primary Performance Endpoint: Rate of All-cause Mortality or Disabling Stroke.
Description: Composite of all-cause mortality or disabling stroke.
Time Frame: 1 year post index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
Participants | 7 | 0

3. Secondary Outcome: Number of Participants With Procedural Success
Description: Defined as absence of procedural mortality AND successful access, delivery of the valve, and retrieval of the delivery system
Time Frame: Procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
Participants | 53 | 12

4. Secondary Outcome: Evaluation of Adverse Event Rates (Descriptive Endpoint)
Description: All-cause mortality, Cardiovascular-related mortality, All Stroke (by severity), Transient Ischemic Attacks (TIA), Myocardial infarction (MI), Coronary obstruction, Minor, Major, and life-threatening bleeding, major vascular complication, access-related non-vascular complication, or cardiac structure complication, acute kidney injury (AKI) stages 1-4, Endocarditis, Clinically significant valve thrombosis.
Time Frame: 30 days post index procedure
Population: All values provided have been rounded to the nearest tenth decimal place.
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
percent
  All-cause mortality | 1.8 | 0.0
  Cardiovascular Mortality | 1.8 | 0.0
  All stroke | 3.5 | 0.0
  Fatal stroke | 0.0 | 0.0
  Stroke with disability | 1.8 | 0.0
  Stroke without disability | 1.8 | 0.0
  TIA | 0.0 | 0.0
  Endocarditis | 0.0 | 0.0
  Clinically significant valve thrombosis | 0.0 | 0.0
  Stage 1 AKI | 0.0 | 7.1
  Stage 2 AKI | 0.0 | 0.0
  Stage 3 AKI | 0.0 | 0.0
  Stage 4 AKI | 0.0 | 7.1
  Type 1 Bleeding | 5.3 | 0.0
  Type 2 Bleeding | 5.3 | 7.1
  Type 3 Bleeding | 0.0 | 21.4
  Type 4 Bleeding | 1.8 | 0.0
  Major Vascular Complication | 1.8 | 21.4
  Major access-related non-vascular complication | 0.0 | 0.0
  Major cardiac structure complication | 1.8 | 0.0
  Myocardial infarction | 0.0 | 0.0
  Coronary obstruction | 0.0 | 0.0

5. Secondary Outcome: Evaluation of Adverse Event Rates (Descriptive Endpoint)
Description: All-cause mortality, Cardiovascular-related mortality, All Stroke (by severity), Transient Ischemic Attacks (TIA), Myocardial infarction (MI), Coronary obstruction, Endocarditis, Clinically significant valve thrombosis.
Time Frame: 1 year post index procedure
Population: Event rates for 1-year follow up and beyond are presented as Kaplan-Meier rates and may not correspond to whole numbers of patients.
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
percent
  All-cause mortality | 10.5 | 0.0
  Cardiovascular Mortality | 7.1 | 0.0
  All stroke | 3.5 | 0.0
  Fatal stroke | 0.0 | 0.0
  Stroke with disability | 1.8 | 0.0
  Stroke without disability | 1.8 | 0.0
  TIA | 1.1 | 0.0
  Endocarditis | 0.0 | 0.0
  Clinically significant valve thrombosis | 0.0 | 0.0
  Myocardial infarction | 1.9 | 0.0
  Coronary obstruction | 4.2 | 0.0

6. Secondary Outcome: Evaluation of Adverse Event Rates (Descriptive Endpoint)
Description: All-cause mortality, Cardiovascular-related mortality, All Stroke (by severity), TIA
Time Frame: 2 years post index procedure
Population: as for outcome 5
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
percent
  All-cause mortality | 12.4 | 15.6
  Cardiovascular Mortality | 9.1 | 0.0
  All stroke | 3.5 | 7.1
  Fatal stroke | 0.0 | 0.0
  Stroke with disability | 1.8 | 7.1
  Stroke without disability | 1.8 | 0.0
  TIA | 1.1 | 0.0
  Endocarditis | 0.0 | 0.0
  Clinically significant valve thrombosis | 0.0 | 0.0

7. Secondary Outcome: Evaluation of Adverse Event Rates (Descriptive Endpoint)
Description: All-cause mortality, Cardiovascular-related mortality, All Stroke (by severity), TIA
Time Frame: 3 years post index procedure
Population: as for outcome 5
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
percent
  All-cause mortality | 24.0 | 15.6
  Cardiovascular Mortality | 13.6 | 0.0
  All stroke | 3.5 | 7.1
  Fatal stroke | 0.0 | 0.0
  Stroke with disability | 1.8 | 7.1
  Stroke without disability | 1.8 | 0.0
  TIA | 1.1 | 0.0
  Endocarditis | 0.0 | 0.0
  Clinically significant valve thrombosis | 0.0 | 0.0

8. Secondary Outcome: Evaluation of Adverse Event Rates (Descriptive Endpoint)
Description: All-cause mortality, Cardiovascular-related mortality, All Stroke (by severity), TIA
Time Frame: 4 years post index procedure
Population: as for outcome 5
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
percent
  All-cause mortality | 38.1 | 15.6
  Cardiovascular Mortality | 19.0 | 0.0
  All stroke | 3.5 | 7.1
  Fatal stroke | 0.0 | 0.0
  Stroke with disability | 1.8 | 7.1
  Stroke without disability | 1.8 | 0.0
  TIA | 1.1 | 0.0
  Endocarditis | 0.0 | 0.0
  Clinically significant valve thrombosis | 0.0 | 0.0

9. Secondary Outcome: Evaluation of Adverse Event Rates (Descriptive Endpoint)
Description: All-cause mortality, Cardiovascular-related mortality, All Stroke (by severity), TIA
Time Frame: 5 years post index procedure
Population: as for outcome 5
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
percent
  All-cause mortality | 45.8 | 15.6
  Cardiovascular Mortality | 19.0 | 0.0
  All stroke | 3.5 | 7.1
  Fatal stroke | 0.0 | 0.0
  Stroke with disability | 1.8 | 7.1
  Stroke without disability | 1.8 | 0.0
  TIA | 1.1 | 0.0
  Endocarditis | 0.0 | 0.0
  Clinically significant valve thrombosis | 0.0 | 0.0

10. Secondary Outcome: Assessment of Clinical Benefit Endpoint - NYHA Class
Description: Change in New York Heart Association (NYHA) functional classification from baseline to 30 days, 1 year, and annually through 5 years.
  The New York Heart Association (NYHA) functional classification is a system used to categorize the severity of heart failure based on the patient's symptoms and functional capacity.
  NYHA Functional Classification
  Class I (No Limitation):
  Class II (Mild Limitation):
  Class III (Moderate Limitation):
  Class IV (Severe Limitation):
  Class I and II are associated with better functional status and quality of life, indicating less severe heart failure. Worse Outcomes: Class III and IV represent more severe heart failure, with significant limitations and increased risk of complications.
Time Frame: 30 days post index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 29 | 8
percent
  Class I | 69.0 | 50.0
  Class II | 24.1 | 37.5
  Class III | 6.9 | 12.5
  Class IV | 0.0 | 0.0

11. Secondary Outcome: Assessment of Clinical Benefit Endpoint - NYHA Class
Description: as for outcome 10
Time Frame: 1 year post index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 29 | 8
percent
  Class I | 54.5 | 40.0
  Class II | 40.9 | 40.0
  Class III | 4.5 | 20.0
  Class IV | 0.0 | 0.0

12. Secondary Outcome: Assessment of Clinical Benefit Endpoint - NYHA Class
Description: as for outcome 10
Time Frame: 2 years post index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 21 | 4
percent
  Class I | 61.9 | 50.0
  Class II | 28.6 | 50.0
  Class III | 9.5 | 0.0
  Class IV | 0.0 | 0.0

13. Secondary Outcome: Assessment of Clinical Benefit Endpoint - NYHA Class
Description: as for outcome 10
Time Frame: 3 years post index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 10 | 3
percent
  Class I | 60.0 | 66.7
  Class II | 10.0 | 0.0
  Class III | 30.0 | 33.3
  Class IV | 0.0 | 0.0

14. Secondary Outcome: Assessment of Clinical Benefit Endpoint - NYHA Class
Description: as for outcome 10
Time Frame: 4 years post index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 4 | 1
percent
  Class I | 75.0 | 100
  Class II | 0.0 | 0.0
  Class III | 25.0 | 0.0
  Class IV | 0.0 | 0.0

15. Secondary Outcome: Assessment of Clinical Benefit Endpoint - NYHA Class
Description: as for outcome 10
Time Frame: 5 years post index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 2 | 1
percent
  Class I | 100.0 | 0.0
  Class II | 0.0 | 0.0
  Class III | 0.0 | 100.0
  Class IV | 0.0 | 0.0

16. Secondary Outcome: Paravalvular Leak as Measured by Core Lab Echocardiography
Description: Paravalvular leak severity was categorized based on echocardiographic criteria, including the size and hemodynamic impact of the leak, as determined by the core lab assessment and categorized under 4 grades: none/trace/trivial; mild; moderate and severe.
Time Frame: 30 Days
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
Participants
  None/trace/trivial: number analyzed (Participants) | 10 | 3
  None/trace/trivial | 10 | 0
  Mild: number analyzed (Participants) | 10 | 3
  Mild | 0 | 0
  Moderate: number analyzed (Participants) | 10 | 3
  Moderate | 0 | 0
  Severe: number analyzed (Participants) | 10 | 3
  Severe | 0 | 0

17. Secondary Outcome: Paravalvular Leak as Measured by Core Lab Echocardiography
Description: as for outcome 16
Time Frame: 1 Year
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
Participants
  None/trace/trivial: number analyzed (Participants) | 6 | 2
  None/trace/trivial | 5 | 2
  Mild: number analyzed (Participants) | 6 | 2
  Mild | 1 | 0
  Moderate: number analyzed (Participants) | 6 | 2
  Moderate | 0 | 0
  Severe: number analyzed (Participants) | 6 | 2
  Severe | 0 | 0

18. Secondary Outcome: Paravalvular Leak as Measured by Core Lab Echocardiography
Description: as for outcome 16
Time Frame: 2 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
Participants
  None/trace/trivial: number analyzed (Participants) | 2 | 2
  None/trace/trivial | 2 | 2
  Mild: number analyzed (Participants) | 2 | 2
  Mild | 0 | 0
  Moderate: number analyzed (Participants) | 2 | 2
  Moderate | 0 | 0
  Severe: number analyzed (Participants) | 2 | 2
  Severe | 0 | 0

19. Secondary Outcome: Paravalvular Leak as Measured by Core Lab Echocardiography
Description: as for outcome 16
Time Frame: 3 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
Participants
  None/trace/trivial: number analyzed (Participants) | 3 | 1
  None/trace/trivial | 2 | 1
  Mild: number analyzed (Participants) | 3 | 1
  Mild | 1 | 0
  Moderate: number analyzed (Participants) | 3 | 1
  Moderate | 0 | 0
  Severe: number analyzed (Participants) | 3 | 1
  Severe | 0 | 0

20. Secondary Outcome: Paravalvular Leak as Measured by Core Lab Echocardiography
Description: as for outcome 16
Time Frame: 4 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
Participants
  None/trace/trivial: number analyzed (Participants) | 1 | 0
  None/trace/trivial | 1 | 0
  Mild: number analyzed (Participants) | 1 | 0
  Mild | 0 | 0
  Moderate: number analyzed (Participants) | 1 | 0
  Moderate | 0 | 0
  Severe: number analyzed (Participants) | 1 | 0
  Severe | 0 | 0

21. Secondary Outcome: Paravalvular Leak as Measured by Core Lab Echocardiography
Description: as for outcome 16
Time Frame: 5 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 57 | 14
Participants
  None/trace/trivial: number analyzed (Participants) | 1 | 1
  None/trace/trivial | 1 | 1
  Mild: number analyzed (Participants) | 1 | 1
  Mild | 0 | 0
  Moderate: number analyzed (Participants) | 1 | 1
  Moderate | 0 | 0
  Severe: number analyzed (Participants) | 1 | 1
  Severe | 0 | 0

22. Secondary Outcome: Mean Transvalvular Gradient as Measured by Core Lab Echocardiography
Description: Echocardiographic examinations were forwarded to the independent echocardiographic core lab MedStar Health Echocardiography Core Laboratory for interpretation. It was the responsibility of each study site to perform the local interpretation of the echocardiogram for clinical assessment.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 19 | 7
mmHg | 13.90 (5.66) | 14.67 (4.82)

23. Secondary Outcome: Mean Transvalvular Gradient as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 19 | 1
mmHg | 11.13 (5.18) | 8.40 (3.58)

24. Secondary Outcome: Mean Transvalvular Gradient as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 2 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 10 | 3
mmHg | 13.49 (6.85) | 11.17 (7.02)

25. Secondary Outcome: Mean Transvalvular Gradient as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 3 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 5 | 4
mmHg | 12.00 (4.78) | 9.05 (4.59)

26. Secondary Outcome: Mean Transvalvular Gradient as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 4 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 1 | 2
mmHg | 19.90 (NA) — Standard Deviation cannot be calculated for one subject. At this time point (4 years), data is only reported for a single subject. | 6.50 (1.84)

27. Secondary Outcome: Mean Transvalvular Gradient as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 5 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 2 | 2
mmHg | 9.15 (2.19) | 14.00 (10.75)

28. Secondary Outcome: Aortic Valve Area as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 15 | 5
cm^2 | 1.47 (0.36) | 1.25 (0.25)

29. Secondary Outcome: Aortic Valve Area as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 1 Year
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 13 | 5
cm^2 | 1.41 (0.32) | 1.82 (0.56)

30. Secondary Outcome: Aortic Valve Area as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 2 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 7 | 3
cm^2 | 1.47 (0.58) | 1.33 (0.12)

31. Secondary Outcome: Aortic Valve Area Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 3 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 3 | 4
cm^2 | 1.63 (0.20) | 1.48 (0.37)

32. Secondary Outcome: Aortic Valve Area as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 4 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 0 | 2
cm^2 |  | 1.72 (0.40)

33. Secondary Outcome: Aortic Valve Area as Measured by Core Lab Echocardiography
Description: as for outcome 22
Time Frame: 5 Years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 1 | 2
cm^2 | 2.09 (NA) — Standard deviation cannot be calculated for one subject. | 1.26 (0.34)

34. Secondary Outcome: New Pacemaker Implant
Description: New permanent pacemaker implantation(PPI), with precision of the indication and the number of days postimplant of the placement of the new permanent pacemaker.
Time Frame: 30 days
Population: Pacemaker implant (PPI) is unique and only applies to a portion of the patients.
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 48 | 14
percent | 4.2 | 0.0

35. Secondary Outcome: New Pacemaker Implant
Description: as for outcome 34
Time Frame: 1 year
Population: Pacemaker implant (PPI) is unique and only applies to a portion of the patients.
Measure: Number; unit: percent
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
Number analyzed (Participants) | 48 | 14
percent | 1.8 | 0.0

ADVERSE EVENTS:
Time Frame: 5 years
Description: Number of subjects as presented in the CSR does not limit the number of times a subject can be counted for another event.
Arm/Group | Primary Analysis Population | Exploratory Registry Arm
All-Cause Mortality (participants affected / at risk) | 16/57 | 2/14
Serious Adverse Events (participants affected / at risk) | 44/57 | 10/14
Other Adverse Events (participants affected / at risk) | 41/57 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Analysis Population (N=57) | Exploratory Registry Arm (N=14)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 2 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 2 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 2
Cardiac Tamponade (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Mitral Valve Incompetence (Cardiac disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 0
Incarcerated Hernia (General disorders) | 0 | 1
Paravalvular Regurgitation (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Covid-19 (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 5 | 1
Pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 3 | 1
Hemoglobin Decreased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Esophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Peripheral Artery Aneurysm (Nervous system disorders) | 1 | 0
Peripheral Artery Occlusion (Nervous system disorders) | 1 | 0
Thrombosis (Nervous system disorders) | 1 | 0
Device Dislocation (Product Issues) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Iliac Artery Rupture (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Analysis Population (N=57) | Exploratory Registry Arm (N=14)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Bundle Branch Block Left (Cardiac disorders) | 4 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Covid-19 (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Delirium (Injury, poisoning and procedural complications) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Intravascular Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Blood Potassium (Investigations) | 0 | 1
Myeloproliferative Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will have the right to publish overall study results. Investigators may publish results from their respective participating site per their discretion but only after the multi-center publication is published or 12 months have passed from the study conclusion without a multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT05002088/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT05002088/SAP_001.pdf